CLINICAL TRIAL: NCT00901134
Title: Multicenter Registry Study With Therapeutic Hypothermia After Cardiac Arrest in Japan
Acronym: J-PULSE-HYPO
Status: Completed | Type: Observational
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Hiroshi Nonogi, Department of Cardiology , National Cardiovascular Center,Japan
Other Study IDs: NCVC-JPULSE-H; UMIN000001935
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Cardiac Arrest
Keywords: therapeutic hypothermia after cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hypothermia: Patients with therapeutic hypothermia after cardiac arrest in hospitals

SUMMARY:
Recently, early defibrillation and cardiopulmonary resuscitation (CPR) for sudden onset of cardiac arrest are advancing, however, survival rate is still very low in the world. Furthermore, post-cardiac arrest brain injury is a common cause of morbidity and mortality after successful resuscitation which is urgent issue to be solved. Therapeutic hypothermia is part of a standardized treatment strategy for comatose survivors of cardiac arrest in the metabolic phase usually about 15 minutes after cardiac arrest. However, the evidences of the efficacy of therapeutic hypothermia are still few. The optimal candidates, temperature, the timing of initiation, the therapeutic windows and the rate for rewarming have not been defined clinically and should be established. The purpose of this research is the improvement in the outcomes for patients with coma after resuscitation from out-of-hospital cardiac arrest using therapeutic hypothermia established from the analysis of multicenter registry data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who remained unconscious after resuscitation from out-of-hospital or inhospital cardiac arrest
* Presented the stable hemodynamics with drug treatments or mechanical supporting system including IABP or PCPS

Exclusion Criteria:

* Patients with:

  * pregnancy
  * acute aortic dissection
  * pulmonary thromboembolism
  * drug poisoning
  * poor daily activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with therapeutic hypothermia after cardiac arrest from 2005 to 2009 in each hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Survival and functional outcome (CPC: Cerebral Performance Categories) | after 3 months

SECONDARY OUTCOMES:
Survival and/or functional outcome | after 24 hours
Survival and/or functional outcome | after 7 days
Survival and/or functional outcome | after one month
Survival and/or functional outcome | at discharge
Survival or functional outcome | after three months

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Nonogi, MD, Principal Investigator — Department of Cardiology, National Cardiovascular Center , Japan
Locations (14):
- Japan (14):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Hiroshima City Hospital, Hiroshima, Hiroshima
  - Sapporo City University Hopistal, Sapporo, Hokaido
  - Kagawa University Hospital, Takamatsu, Kagawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka Police Hospital, Osaka, Osaka
  - Sumitomo Hospital, Osaka, Osaka
  - National Cardiovascular Center, Suita, Osaka
  - Osaka Saiseikai Senri Hospital, Suita, Osaka
  - Osaka Mishima Emergency Critical Care Center, Takatsuki, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - Nihon University Surugadai Hospital, Tokyo, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi

REFERENCES:
- [Result] Yokoyama H, Nagao K, Hase M, Tahara Y, Hazui H, Arimoto H, Kashiwase K, Sawano H, Yasuga Y, Kuroda Y, Kasaoka S, Shirai S, Yonemoto N, Nonogi H; J-PULSE-Hypo Investigators. Impact of therapeutic hypothermia in the treatment of patients with out-of-hospital cardiac arrest from the J-PULSE-HYPO study registry. Circ J. 2011;75(5):1063-70. doi: 10.1253/circj.cj-11-0137. Epub 2011 Apr 7. PMID 21471669
- [Derived] Soga T, Nagao K, Sawano H, Yokoyama H, Tahara Y, Hase M, Otani T, Shirai S, Hazui H, Arimoto H, Kashiwase K, Kasaoka S, Motomura T, Kuroda Y, Yasuga Y, Yonemoto N, Nonogi H; J-PULSE-Hypo Investigators. Neurological benefit of therapeutic hypothermia following return of spontaneous circulation for out-of-hospital non-shockable cardiac arrest. Circ J. 2012;76(11):2579-85. doi: 10.1253/circj.cj-12-0448. Epub 2012 Jul 20. PMID 22813874
- See also: Related Info — http://j-pulse.umin.jp/